CLINICAL TRIAL: NCT06784427
Title: Normal Reference Values for 3T Cardiac Parametric Mapping
Acronym: NORMAP3T
Status: Completed | Type: Observational
Sponsor: IRCCS Azienda Ospedaliero-Universitaria di Bologna (Other)
Responsible Party: Sponsor
Other Study IDs: NORMAP3T
Record Dates: First submitted 2025-01-09; First posted 2025-01-20 (Actual); Last update posted 2025-01-20 (Actual); Status verified 2024-11

CONDITIONS: Cardiac Imaging; Cardiac Imaging Techniques

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This is a study non-randomised and uncontrolled cross-sectional experimental/interventional study.

Consecutive subjects will be enrolled healthy, volunteer subjects to undergo a Cardio-RM examination on the new 3T MRI equipment.

The Cardio-RM examination to which they will undergo: does NOT involve the administration of contrast medium involves the performance of certain preliminary 'localisation' sequences.

Following the execution of the investigation the investigators will use the post-processing workstations to analyse the parametric sequences and extract the T1 and T2 values of the myocardium.

To minimise bias, two different investigators different experimenters independently evaluate the sequences, in order to assess inter-observer agreement; furthermore, to assess the stability of the acquisition of these sequences, temperature and humidity will be measured of the MRI room for each survey performed.

DETAILED DESCRIPTION:
Cardiac MRI represents the gold standard for the in vivo differentiation of various types of cardiomyopathies, thanks to its ability to characterize tissue. Through specific parametric mapping sequences, cardiac MRI allows not only the identification but also the quantification of both focal and diffuse alterations that cannot be assessed with other techniques. These sequences enable the direct measurement of relaxation times T1 (spin-lattice) and T2 (spin-spin), expressed in milliseconds, thus providing the ability to differentiate various tissue alterations (e.g., inflammation, ischemia, edema, and fibrosis).

The usefulness of T1 mapping sequences in analyzing certain cardiomyopathies, such as cardiac involvement in Anderson-Fabry disease, amyloidosis, and hemochromatosis, is well-documented in the literature. Similarly, T2 mapping sequences are valuable for evaluating inflammatory processes and myocarditis. Parametric sequences are also used to assess rejection phenomena in patients undergoing cardiac transplantation and play a crucial role in evaluating various cardiomyopathies in their end-stage phases.

Despite the broad and promising applications of these sequences as reported in the literature, certain challenges persist in their use. Specifically, the normal values for these sequences vary depending on the type of sequence and the specific MRI equipment employed. In our department, these sequences have been routinely used in clinical practice with a 1.5T MRI machine, for which the normal values have already been established and documented. With the recent installation of a new 3T MRI system, it is therefore necessary to determine the normal values of parametric sequences in healthy subjects to enable their use in routine clinical practice and for research purposes involving patients with various types of cardiomyopathies.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy volunteers with a negative history of established cardiac disease
2. 20-70 years old
3. Acquisition of informed consent

Exclusion Criteria:

1. Positive family history of known cardiomyopathies, sudden cardiac death
2. Taking specific chronic therapy for diabetes and hypertension with ≥ 2 drugs and/or
3. Cardio-vascular risk factors: obesity, hypertension on ≥ 2 drugs, smoking (>10 cigarettes/day)
4. Competitive sports subjects or athletes (defined as >9 hours of sports activity/week)
5. Pregnant women
6. Claustrophobic subjects
7. Other absolute contraindications to MRI
8. Subjects with a relationship of direct/indirect subordination from the Radiology Unit, IRCCS - Azienda Ospedaliero Universitaria di Bologna Policlinico S. Orsola-Malpighi

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Healthy volunteers with a negative history of established cardiac disease
Sampling Method: Non-Probability Sample
Enrollment: 143 (Actual)
Dates: Start 2023-09-26 (Actual); Primary Completion 2024-04-19 (Actual); Study Completion 2024-04-19 (Actual)

PRIMARY OUTCOMES:
Normal T1 mapping values at 3T | Form date of examination until 3 months
  To establish the normal values of the T1 mapping with a 3T MRI in healthy subjects, measuring the mean and standard deviation of the values obtained from the specific sequence
Normal T2 mapping values at 3T | Form date of examination until 3 months
  To establish the normal values of the T2 mapping with a 3T MRI in healthy subjects, measuring the mean and standard deviation of the values obtained from the specific sequence

CONTACTS AND LOCATIONS:
Overall Officials: Edoardo Rasciti, MD, Principal Investigator — IRCCS Azienda Ospedaliero-Universitaria di Bologna
Locations (1):
- IRCCS Azienda Ospedaliero-Universitaria di Bologna, Bologna, Italy